CLINICAL TRIAL: NCT05858359
Title: Contextualized Neuropsychological Rehabilitation for CNS Cancer Survivors: The "I'm Aware: Patients and Carers Together" (ImPACT) Program"
Brief Title: Contextualized Neuropsychological Rehabilitation for CNS Cancer Survivors: The ImPACT Program
Acronym: ImPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Lisa Maria Wu, Associate Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ImPACT Adult
Record Dates: First submitted 2023-05-01; First posted 2023-05-15 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Brain Cancer; Cognitive Impairment
Keywords: Brain Cancer; Brain Tumor; Cognitive Impairment; Neurobehavioral Impairment; Neuropsychological Rehabilitation
MeSH Terms: conditions — Brain Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized waitlist controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ImPACT program (Experimental): The ImPACT program consists of 8 weekly 1-hour sessions with homework between sessions.
  Interventions: Behavioral: ImPACT program
- Waitlist (No Intervention): Waitlist control

INTERVENTIONS:
Behavioral: ImPACT program — During the ImPACT program, the brain cancer survivor and a carer collaborate on:
  1. Becoming aware of the patient's core strengths and difficulties
  2. Helping the patient to be optimally responsive to the guidance of the carer, and
  3. Creating compensatory strategies to respond to real-world manifestations of the patient's difficulties and helping the patient implement these strategies at home.
  Arms: ImPACT program

SUMMARY:
The aim of the present randomized-controlled study is to evaluate the feasibility, acceptability, and preliminary efficacy of a novel, context-sensitive neuropsychological rehabilitation intervention for brain cancer survivors.

DETAILED DESCRIPTION:
Cognitive impairment is the most common late effect in brain cancer survivors, with profound negative effects on quality of life, work ability, and socioeconomic outcomes. Still, there is no gold standard approach to treating cognitive impairment in brain cancer survivors. Furthermore, there is a dearth of research on interventions to treat cognitive impairment in brain cancer survivors, and the relatively few studied interventions have proven limited effects. Arguably, four key elements are missing from a majority of studied interventions:1) transfer of learning to real-world functional outcomes, 2) awareness training to enhance compensatory strategy use, 3) inclusion of carers that could enhance transfer of learning to the home, and 4) recognition of the inter-related nature of cognitive, neurobehavioral, and psychological functions.

The "I'M aware: Patients and Carers Together (ImPACT)" program is a novel, context-sensitive neuropsychological rehabilitation intervention that targets the above mentioned missing elements in previous rehabilitation efforts. The present feasibility randomized-controlled study aims to evaluate the feasibility, acceptability, and preliminary efficacy of this program in brain cancer survivors with cognitive impairment in preparation for a subsequent large-scale randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of brain cancer
* Completed primary treatment at least 6 months ago
* Medically stable
* Speaks and understand Danish
* Living with a carer aged 18 or over, who also speaks and understands Danish and consents to participate in the study alongside the patient

Exclusion Criteria:

• Confounding diagnosed or suspected psychiatric or medical condition unrelated to the cancer or its treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Self-reported cognitive functioning | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Patients Assessment of Own Functioning Inventory (PAOFI). 33 items: answer format range 1-6; total score range: 0-33. Higher score indicates more impairment.
Carer-reported cognitive functioning | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Patients Assessment of Own Functioning Inventory (PAOFI) modified to informant version. 33 items: answer format range 1-6; total score range: 0-33. Higher score indicates more impairment.
Self-reported neurobehavioral functioning | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The self-report version of the Frontal Systems Behavior Scale (FrSBe). 46 items: answer format range 1-5; total score range: 46-230. Higher score indicates more impairment.
Carer-reported neurobehavioral functioning | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The carer-report version of the Frontal Systems Behavior Scale (FrSBe). 46 items: answer format range 1-5; total score range: 46-230. Higher score indicates more impairment.

SECONDARY OUTCOMES:
Self-reported cognitive functioning | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Patients Assessment of Own Functioning Inventory (PAOFI). 33 items: answer format range 1-6; total score range: 0-33. Higher score indicates more impairment.
Carer-reported cognitive functioning | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Patients Assessment of Own Functioning Inventory (PAOFI) modified to informant version. 33 items: answer format range 1-6; total score range: 0-33. Higher score indicates more impairment.
Self-reported neurobehavioral functioning | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The self-report version of the Frontal Systems Behavior Scale (FrSBe). 46 items: answer format range 1-5; total score range: 46-230. Higher score indicates more impairment.
Carer-reported neurobehavioral functioning | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The carer-report version of the Frontal Systems Behavior Scale (FrSBe). 46 items: answer format range 1-5; total score range: 46-230. Higher score indicates more impairment.
Objective cognitive functioning (Neuropsychological tests; Patient only) | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  Global composite z-score based on the HVLT-R; Trail-making tests A and B; WAIS-IV Coding, Digit Span, Verbal Fluency; Conner's Continuous Performance Test III.
Objective cognitive functioning (Neuropsychological tests; Patient only) | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  Global composite z-score based on the HVLT-R; Trail-making tests A and B; WAIS-IV Coding, Digit Span, Verbal Fluency; Conner's Continuous Performance Test III.
Premorbid intellectual functioning (Patient only) | Baseline (T1)
  WAIS-IV Information subtest. 26 items; answer format range 0-1; total score range: 0-26. Higher score indicates higher premorbid intellectual functioning.
Self-reported fatigue | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Functional Assessment of Chronic Illness Therapy-Fatigue scale (FACIT-Fatigue). 13 items: answer format range 0-4; total score range: 0-52. Lower score indicates more fatigue.
Carer-reported fatigue | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Functional Assessment of Chronic Illness Therapy-Fatigue scale (FACIT-Fatigue) modified to informant version. 13 items: answer format range 0-4; total score range: 0-52. Lower score indicates more fatigue.
Self-reported fatigue | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Functional Assessment of Chronic Illness Therapy-Fatigue scale (FACIT-Fatigue). 13 items: answer format range 0-4; total score range: 0-52. Lower score indicates more fatigue.
Carer-reported fatigue | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Functional Assessment of Chronic Illness Therapy-Fatigue scale (FACIT-Fatigue) modified to informant version. 13 items: answer format range 0-4; total score range: 0-52. Lower score indicates more fatigue.
Self-reported mental fatigue | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Mental Fatigue Scale (MFS). 15 items: answer format range 0-3; total score range: 0-45. Higher score indicates more mental fatigue.
Carer-reported mental fatigue | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Mental Fatigue Scale (MFS) modified to informant version. 15 items: answer format range 0-3; total score range: 0-45. Higher score indicates more mental fatigue.
Self-reported mental fatigue | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Mental Fatigue Scale (MFS). 15 items: answer format range 0-3; total score range: 0-45. Higher score indicates more mental fatigue.
Carer-reported mental fatigue | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Mental Fatigue Scale (MFS) modified to informant version. 15 items: answer format range 0-3; total score range: 0-45. Higher score indicates more mental fatigue.
Depression (patient only) | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Center for Epidemiologic Studies Depression Scale (CESD). 20 items: answer format range 0-3; total score range: 0-60. Higher score indicates more depression.
Depression (patient only) | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Center for Epidemiologic Studies Depression Scale (CESD). 20 items: answer format range 0-3; total score range: 0-60. Higher score indicates more depression.
Self-reported health-related quality of life | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Functional Assessment of Cancer Therapy-Brain (FACT-Br). 50 items; answer format range 0-4; total score range: 0-200. Higher score indicates better health-related quality of life.
Carer-reported health-related quality of life | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Functional Assessment of Cancer Therapy-Brain (FACT-Br) modified to informant version. 50 items; answer format range 0-4; total score range: 0-200. Higher score indicates better health-related quality of life.
Self-reported health-related quality of life | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Functional Assessment of Cancer Therapy-Brain (FACT-Br). 50 items; answer format range 0-4; total score range: 0-200. Higher score indicates better health-related quality of life.
Carer-reported health-related quality of life | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Functional Assessment of Cancer Therapy-Brain (FACT-Br) modified to informant version. 50 items; answer format range 0-4; total score range: 0-200. Higher score indicates better health-related quality of life.
Self-reported community integration | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The self-report version of the Community Integration Questionnaire Revised (CIQ-R). 18 items: answer format range 0-2; total score range: 0-35. Higher score indicates more community integration.
Carer-reported community integration | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The carer-report version of the Community Integration Questionnaire Revised (CIQ-R). 18 items: answer format range 0-2; total score range: 0-35. Higher score indicates more community integration.
Self-reported community integration | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The self-report version of the Community Integration Questionnaire Revised (CIQ-R). 18 items: answer format range 0-2; total score range: 0-35. Higher score indicates more community integration.
Carer-reported community integration | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The self-report version of the Community Integration Questionnaire Revised (CIQ-R). 18 items: answer format range 0-2; total score range: 0-35. Higher score indicates more community integration.
Insomnia | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Insomnia Severity Index (ISI). 7 items; answer format range: 0-4; total score range: 0-28. Higher score indicates more insomnia.
Insomnia | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Insomnia Severity Index (ISI). 7 items; answer format range: 0-4; total score range: 0-28. Higher score indicates more insomnia.
Self-reported participant satisfaction | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Client Satisfaction Questionnaire (CSQ-8). 8 items: answer format range 1-4; total score range: 8-32. Higher score indicates better satisfaction.
Carer-reported participant satisfaction | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The Client Satisfaction Questionnaire (CSQ-8). 8 items: answer format range 1-4; total score range: 8-32. Higher score indicates better satisfaction.
Self-reported participant satisfaction | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Client Satisfaction Questionnaire (CSQ-8). 8 items: answer format range 1-4; total score range: 8-32. Higher score indicates better satisfaction.
Carer-reported participant satisfaction | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The Client Satisfaction Questionnaire (CSQ-8). 8 items: answer format range 1-4; total score range: 8-32. Higher score indicates better satisfaction.
Self-reported participant motivation | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The 7-item interest/enjoyment subscale of the Intrinsic Motivation Inventory (IMI). 7 items: answer format range 1-7; total score range: 1-7. Higher score indicates more motivation.
Carer-reported participant motivation | Baseline (T1) to after last session (approximately 8 weeks later: Post-intervention, T3)
  The 7-item interest/enjoyment subscale of the Intrinsic Motivation Inventory (IMI). 7 items: answer format range 1-7; total score range: 1-7. Higher score indicates more motivation.
Self-reported participant motivation | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The 7-item interest/enjoyment subscale of the Intrinsic Motivation Inventory (IMI). 7 items: answer format range 1-7; total score range: 1-7. Higher score indicates more motivation.
Carer-reported participant motivation | Baseline (T1) to 8 week after post-intervention (approximately 16 weeks later: Follow-up, T4)]
  The 7-item interest/enjoyment subscale of the Intrinsic Motivation Inventory (IMI). 7 items: answer format range 1-7; total score range: 1-7. Higher score indicates more motivation.

OTHER OUTCOMES:
Qualitative Interviews | 8 weeks after post-intervention (approximately 16 weeks after Baseline assessment (T1): Follow-up, T4)
  Following the T4 assessment, participants included in the intervention arm will be invited to participate in a 30-minutes semi-structured, audio recorded interview.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Wu, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No